CLINICAL TRIAL: NCT03585816
Title: Qualitative Assessment of the Composition of the Exhaust Gas of Pneumoperitoneum During Laparoscopic Surgery: Prospective Gas Chromatographic Study
Brief Title: Composition of the Exhaust Gas of Pneumoperitoneum During Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: Gas-chromato-P.Diemunsch
Record Dates: First submitted 2018-06-20; First posted 2018-07-13 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2018-06

CONDITIONS: Pneumoperitoneum
Keywords: Pneumoperitoneum; Exhaust gas; chromatographic study; Nitrous oxide; Nitrogen dioxide
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research aims to study the composition of the peritoneal exhaust gas during laparoscopic surgery to detect and possibly quantify the presence of air and / or N2O. This purely descriptive work is part of other experimental work that the investigators have already published.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient who will benefit from a laparoscopic surgery at Strasbourg University Hospitals
* Patient who has consented to the use of her medical data for research purposes.

Exclusion Criteria:

- Refusal of the patient to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient who will benefit from a laparoscopic surgery at Strasbourg University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
to quantify the composition of the exhaust gas of pneumoperitoneum during laparoscopic surgery by gas chromatography | 1 day after laparoscopic surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Service d' Anesthésie Réanimation Chirurgicale, Strasbourg, France